CLINICAL TRIAL: NCT01481519
Title: A Randomized, Double-Masked Trial of Topical Dexamethasone 0.1%/Povidone-iodine 0.4% Versus Artificial Tears for Treatment of Viral Conjunctivitis
Brief Title: A Trial of Topical Dexamethasone Versus Artificial Tears for Treatment of Viral Conjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Joao Paulo Felix, Dr., University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0664.0.146.000-11
Record Dates: First submitted 2011-11-13; First posted 2011-11-29 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Viral Conjunctivitis
Keywords: Conjunctivitis; Ocular diseases; Artificial tears
MeSH Terms: conditions — Conjunctivitis, Viral; Conjunctivitis | interventions — Dexamethasone; Lubricant Eye Drops

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dexamethasone 0.1%/povidone-iodine 0.4% (Active Comparator): Patients were instructed to put one drop into each symptomatic eye four times daily for 7 days.
  Interventions: Drug: dexamethasone 0.1%/povidone-iodine 0.4%
- artificial tears (Placebo Comparator): Patients were instructed to put one drop into each symptomatic eye four times daily for 7 days.
  Interventions: Drug: Artificial Tears

INTERVENTIONS:
Drug: dexamethasone 0.1%/povidone-iodine 0.4% — dexamethasone 0.1%/povidone-iodine 0.4%
  Other Names: Dexamethasone / Iodo - povidone
  Arms: dexamethasone 0.1%/povidone-iodine 0.4%
Drug: Artificial Tears — artificial tears 1 drop, 4 times per day
  Arms: artificial tears

SUMMARY:
Viral conjunctivitis causes redness, tearing, swelling, and irritation of the eyes that typically lasts from 1 to 3 weeks. Current management of this condition focuses on supportive care while the viral infection completes its course and resolves. However, many patients still experience substantial discomfort despite standard treatments, and, given the disproportionate morbidity and potential economic impact associated with an outbreak of infective conjunctivitis, a therapeutic agent that reduces clinical symptoms of and minimizes shedding of infectious virus would be desirable.

Povidone-iodine is an antiseptic extensively used in preparation for general surgery, ophthalmic purposes, and laboratory disinfection. Dilute povidone-iodine solutions inhibit numerous viruses, bacteria, fungi, and some other parasites. Low cost, effectiveness, and lack of microbial resistance make povidone-iodine an appealing drug to treat ocular infections, especially in developing countries. Previously studies showed that povidone-iodine is a potential option to reduce contagiousness in cases of adenoviral infections. Dexamethasone 0.1%/povidone-iodine 0.4% it is a mixture containing a steroid and antiseptic is promising as a suitable therapeutic agent for the treatment of EKC. A small, prospective, open-label, single-armed clinical trial of dexamethasone 0.1%/povidone-iodine 0.4% administration in humans with symptoms of acute conjunctivitis who tested positive for adenoviral antigen was therapeutically successful. In other study, dexamethasone 0.1%/povidone-iodine 0.4% combination markedly lowered the viral concentration and improved the manifestations of the disease.

So, the favorable human data in combination with in vivo results provide a strong impetus for a human phase III clinical trial to test the efficacy of this drug in a larger group and also to evaluate complete safety to properly establish the therapeutic benefit versus adverse effect for these reasons, the investigators chose to study the efficacy of dexamethasone 0.1%/povidone-iodine 0.4% in treating the symptoms and signs of viral conjunctivitis. The administration of dexamethasone 0.1%/povidone-iodine 0.4% can be a secure, tolerable and affective treatment to inflammatory and infective component of acute viral conjunctivitis.

DETAILED DESCRIPTION:
Patients who met the study criteria and who agreed to participate in the study were randomly assigned to receive either dexamethasone 0.1%/povidone-iodine 0.4% or artificial tears. Sealed, randomly numbered opaque manila envelopes containing unlabeled bottles of either dexamethasone 0.1%/povidone-iodine 0.4% or artificial tears were given to the patient. Patients were instructed to put one drop into each symptomatic eye four times daily for 7 days. The identity of the drops was masked to both the investigators and patients until the study was closed. At the end of the study, the code for the randomization scheme was obtained. This study was approved by an ethics committee linked to the Institution of origin, and written informed consent was obtained from all patients.

Patients were evaluated at baseline and were asked to return either 5, 10 and 30 days later for a follow-up evaluation. The principal efficacy variables were six symptoms of viral conjunctivitis: overall discomfort, itching, foreign body sensation, tearing, redness, and lid swelling. Four signs of viral conjunctivitis were also evaluated: conjunctival injection, conjunctival chemosis, conjunctival mucus, and lid edema.

Each of the symptoms was rated by the patient at presentation and at follow-up on a 4 point scale: none (0), mild (1), moderate (2), or severe (3). In addition, each patient was asked to report their opinion on the usefulness of the treatment in relieving their symptoms on a 4-point scale: did not help (0), unsure (1), think it helped (2), and sure it helped (3).

ELIGIBILITY:
Inclusion Criteria:

* unilateral or asymmetric conjunctivitis,
* follicles on the inferior tarsal conjunctiva,
* preauricular lymphadenopathy,
* an associated upper respiratory infection or
* recent contact with a person with a red eye

Exclusion Criteria:

* history of seasonal allergic conjunctivitis,
* use of ocular medication after the beginning of symptoms,
* contact lens wear,
* history of herpetic eye disease,
* history of ocular surgery,
* history of chronic ocular disease other than refractive error,
* allergy to iodo, pregnancy,
* age less than 18 years,
* bleeding disorder,
* glaucoma,
* significant blepharitis or dry eyes on slit lamp examination,
* purulent ocular discharge,
* corneal epithelial staining with fluorescein, or
* intraocular inflammation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Conjunctival injection | Day 5 of symptom
  Patient´s information.
  Each of the symptoms was rated by the patient at presentation and at follow-up on a 4 point scale: none (0), mild (1), moderate (2), or severe (3).

SECONDARY OUTCOMES:
Conjunctival chemosis | Day 10 of symptom
  Patient´s information.
  Each of the symptoms was rated by the patient at presentation and at follow-up on a 4 point scale: none (0), mild (1), moderate (2), or severe (3).
Conjunctival chemosis | Day 30 of symptom
  Patient´s information.
  Each of the symptoms was rated by the patient at presentation and at follow-up on a 4 point scale: none (0), mild (1), moderate (2), or severe (3).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Pessoa C Lira, Study Chair — University of Campinas
Locations (1):
- University of Campinas, Campinas, São Paulo, Brazil

REFERENCES:
- [Background] Sambursky RP, Fram N, Cohen EJ. The prevalence of adenoviral conjunctivitis at the Wills Eye Hospital Emergency Room. Optometry. 2007 May;78(5):236-9. doi: 10.1016/j.optm.2006.11.012. PMID 17478342
- [Background] O'Brien TP, Jeng BH, McDonald M, Raizman MB. Acute conjunctivitis: truth and misconceptions. Curr Med Res Opin. 2009 Aug;25(8):1953-61. doi: 10.1185/03007990903038269. PMID 19552618
- [Background] Romanowski EG, Roba LA, Wiley L, Araullo-Cruz T, Gordon YJ. The effects of corticosteroids of adenoviral replication. Arch Ophthalmol. 1996 May;114(5):581-5. doi: 10.1001/archopht.1996.01100130573014. PMID 8619769
- [Result] 2. Cullom RD Jr, Chang B, eds. The Wills Eye Manual: Office and Emergency Room Diagnosis and Treatment of Eye Diseases, 2nd ed. Philadelphia: J.B. Lippincott, 1994; chap 5.
- See also: Related Info — http://www.fcm.unicamp.br